CLINICAL TRIAL: NCT05941182
Title: Co-designing and Evaluating a Real-world Implementation Model for Remote Consultation with Vision Self-testing. the ReVise Study.
Brief Title: Co-designing and Evaluating a Real-world Implementation Model for Remote Consultation with Vision Self-testing.
Acronym: ReVise
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); University of East Anglia (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Louise Allen, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A096658
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ophthalmic Disorders
Keywords: Remote consultation; visual acuity testing; self-testing applications; home-testing applications
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient participants: Participants who have been assigned to remote consultation follow up following a face-to-face appointment by their clinician.
  Online Perceived Attributes of eHealth Technology online questionnaire before and after the remote consultation.
  Interventions: Other: online questionnaires
- Staff participants: Medical and administrative eye clinic staff at participating centres. Normalisation process (NOMAD) online questionnaire before and after the implementation period.
  Interventions: Other: online questionnaires

INTERVENTIONS:
Other: online questionnaires — Before and after online questionnaires

SUMMARY:
This study aims to involve the public, patients and National Health Service (NHS) staff in co-designing a scalable, inclusive and sustainable implementation model for ophthalmic remote consultation with vision self-testing (the intervention). The main study questions are:

What are the barriers to uptake of the intervention and how can these be mitigated by the design of the implementation model.

How do implementation outcome measures compare before and after real world application of the model.

DETAILED DESCRIPTION:
Background: Increasing demand for hospital eyecare and limited resources makes improved uptake of remote consultation essential. Unsupported workflows and the lack of an accurate visual acuity (VA) assessment are recognised factors limiting its uptake by ophthalmologists. Difficulties with accessing and trusting technology are widely reported barriers for patients. A novel implementation model of remote consultation with vision selftesting (using the DigiVis app in this study) which is co-designed with stakeholders could support and promote its use.

Methods: This mixed methodology, highly pragmatic study will take place in three large NHS eye departments (in Cambridge, Peterborough and Manchester) with high levels of age, ethnic, cultural and socio-economic diversity. Qualitative and quantitative data from semi-structured interviews, ethnographic field notes in the community and the Planning and Evaluating Remote Consultation Services (PERCS) framework in hospital-based patient and staff focus groups will identify implementation challenges. An implementation model to mitigate these challenges will be co-designed with stakeholders and put into operation. Patients will be allocated to the intervention pathway at their clinician's discretion and with their implied agreement in accepting the appointment.

Implementation and service outcomes will be assessed using the Practical, Robust, Implementation and Sustainability Model of the Reach Effectiveness Adoption Implementation Maintenance (PRISM RE-AIM) framework before, during and after 14 months of operation, enabling adaptation of the model.

Online questionnaires of approximately 100 patients assigned to the intervention by their clinician, will enable quantitative analysis of change in patients' perceived attributes of the e-health innovation scores before and after its use. Online questionnaires will enable quantitative changes in the Normalisation Process (NoMAD) scores of approximately 100 staff before and after implementation of the co-deisgned model to be analysed by descriptive statistics.

The optimised implementation model for the intervention, when scaled up, could reach over 3 million patients a year and alleviate some of the pressures on United Kingdom (UK) ophthalmology services. Dissemination of the model and toolkit via websites, publications and presentations to patients, clinicians, service managers and policy makers will supportthe adoption of remote consultations using self-assessment apps, like DigiVis. This could not only improve patient care in the NHS but improve access to eyecare and vision screening for rural communities internationally.

ELIGIBILITY:
Inclusion Criteria:

* Patients 4 years and older scheduled by their clinician for a follow up remote eye clinic consultation following an initial face-to face consultation.

Exclusion Criteria:

-Patients refusing remote consultation or converted to a face-to-face appointment following scheduling.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients will reflect the diversity of the eye clinic population in terms of gender, age, social deprivation, ethnicity and sub-specialty eye condition.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported perceived attributes of e-health innovation score | 30 months
  Change in the perceived attributes of e-health innovation score before and after experiencing remote consultation and self-testing of vision. This questionnaire results in a summated score for each patient with a minimum of 0 and a maximum of 100. Change in overall score before and after the remote consultation will be calculated for each patient and a mean change in score calculated. A higher magnitude positive change in score reflects an improved perception of the technology after the experience.
Change in staff reported normalisation measure of the technology (NoMAD) score | 30 months
  Change in the NoMAD score before and after implementation of the remote consultation and self-testing of vision.This questionnaire results in a summated score for each patient with a minimum of 0 and a maximum of 100. Change in overall score before and after service implementation the remote consultation will be calculated for each member of staff and a mean change in score calculated. A higher magnitude positive change in score reflects improved normalisation and acceptance of the technology after implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Allen, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospital NHS Trust, Cambridge, Cambridgeshire
  - Manchester University Hospitals NHS Trust, Manchester